CLINICAL TRIAL: NCT07354750
Title: Effect of Parasternal Plane Block on Intraoperative Nociception in Pediatric Cardiac Surgery
Brief Title: Effect of Parasternal Plane Block on Intraoperative Nociception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEŞH-EK-2026-010
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Median Sternotomy; Pain Management
Keywords: Median Sternotomy; Parasternal Plane Block
MeSH Terms: conditions — Agnosia | interventions — Population Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parasternal Plane Block (Active Comparator): Patients in this arm will receive standard general anesthesia combined with ultrasound-guided bilateral parasternal plane block. The block will be performed after induction of anesthesia using 0.25% bupivacaine, with a total dose of 1.5 mg/kg, administered in equal volumes to both sides. Intraoperative nociception will be monitored using the Pain Index Monitor (PAM).
  Interventions: Procedure: Parasternal Plane Block
- Group without peripheral nerve block (Active Comparator): Patients in this arm will receive standard general anesthesia without regional anesthesia techniques. Intraoperative nociception will be monitored using the Pain Index Monitor (PAM).
  Interventions: Procedure: Group without peripheral nerve block

INTERVENTIONS:
Procedure: Parasternal Plane Block — Ultrasound-guided bilateral parasternal plane block will be performed after induction of general anesthesia. The block will be performed after induction of anesthesia using 0.25% bupivacaine, with a total dose of 1.5 mg/kg, administered in equal volumes to both sides. The procedure will be carried out by experienced anesthesiologists under sterile conditions.
  Arms: Parasternal Plane Block
Procedure: Group without peripheral nerve block — Patients assigned to this group will undergo the surgical procedure under standard general anesthesia without the use of any peripheral nerve block techniques.
  Arms: Group without peripheral nerve block

SUMMARY:
Effective pain control during pediatric cardiac surgery remains a major clinical challenge, particularly in procedures involving median sternotomy, which is associated with intense nociceptive stimulation. Inadequate intraoperative analgesia may lead to increased opioid requirements, hemodynamic instability, delayed extubation, and prolonged intensive care unit stay. Objective monitoring of nociception may provide valuable information beyond conventional hemodynamic parameters in this vulnerable population.

This prospective randomized controlled study aims to evaluate the effect of ultrasound-guided parasternal plane block on intraoperative nociception in pediatric patients undergoing cardiac surgery with median sternotomy. Intraoperative nociception will be objectively assessed using the Pain Index Monitor (PAM), based on skin conductance measurements.

The results of this study are expected to provide objective evidence regarding the efficacy of parasternal plane block in attenuating nociceptive responses during pediatric cardiac surgery and to support the integration of regional anesthesia techniques and objective nociception monitoring into perioperative pain management strategies for children.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 7 years
* Scheduled for elective congenital cardiac surgery
* Planned median sternotomy
* American Society of Anesthesiologists (ASA) physical status II-III
* Hemodynamically stable preoperative condition
* Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Emergency surgery or redo sternotomy
* Age <6 months or >7 years
* ASA physical status I or >III
* Severe neurological disorders preventing reliable application of behavioral pain scales
* Failure to obtain written informed consent from a parent or legal guardian

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Intraoperative PAM Pain Index | While administering anesthesia during the procedure/surgery
  Comparison of intraoperative Pain Index Monitor (PAM) values between groups in pediatric patients undergoing cardiac surgery via median sternotomy. PAM Pain Index values will be recorded at predefined time points, including after induction of anesthesia, after block performance, at skin incision, during sternotomy, and during sternum closure.

SECONDARY OUTCOMES:
Intraoperative Remifentanil Consumption | While administering anesthesia during the procedure/surgery
  Comparison of total intraoperative remifentanil consumption between groups
Extubation Time | On the operation day
  Comparison of the time from the end of surgery to tracheal extubation between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)